CLINICAL TRIAL: NCT04685447
Title: Inflammatory Cytokine Profile in Maintenance Hemodialysis Patients Affected by COVID-19: Effects of 2 Different Dialysis Strategies
Brief Title: Effects of Different Dialysis Strategies on Inflammation in COVID-19 Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Collaborators: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Pasquale Esposito, Professor, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CER Liguria: 135/20
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Hemodialysis Complication; Inflammatory Response
Keywords: Hemodialysis; Covid19; Inflammation
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expanded Hemodialysis (Experimental): Hemodialysis modality performed by using a medium cut-off membrane
  Interventions: Procedure: Expanded Hemodialysis for Covid19 maintenance hemodialysis patients
- Protein-leaking hemodialysis (Experimental): Hemodialysis modality performed by using a membrane with accentuated absorption capacities.
  Interventions: Procedure: Hemodialysis by protein-leaking dialyzer for Covid19 maintenance hemodialysis patients

INTERVENTIONS:
Procedure: Expanded Hemodialysis for Covid19 maintenance hemodialysis patients — After Covid19 diagnosis participants are randomized to receive Expanded Hemodialysis for two weeks
  Arms: Expanded Hemodialysis
Procedure: Hemodialysis by protein-leaking dialyzer for Covid19 maintenance hemodialysis patients — After Covid19 diagnosis participants are randomized to receive hemodialysis by protein-leaking dialyzer for two weeks
  Arms: Protein-leaking hemodialysis

SUMMARY:
In the course of Coronavirus Disease-19 (COVID-19) uncontrolled inflammation has been related to disease severity and unfavorable outcomes.

Here, the investigators study the longitudinal changes of pro- and anti-inflammatory markers in a population of patients undergoing maintenance hemodialysis (HD) affected by COVID-19, evaluating the potential modulating effects of two different dialysis approaches

DETAILED DESCRIPTION:
For this prospective randomized study, the investigators recruit maintenance hemodialysis patients with confirmed COVID-19 infection. After diagnosis, the patients are randomized to two different dialysis modalities, expanded HD (HDx), performed by use of a medium cut-off membrane, and standard treatment based on the use of a protein-leaking dialyzer (PLD).

The investigators collect clinical and laboratory data, including circulating pre and post-dialysis levels of interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), soluble TLR4 (sTLR4), and interferon-gamma (IFN-g). Samples are collected at diagnosis (T0), and one and two weeks after the diagnosis (T7 and T14, respectively). Moreover, lymphocyte and immune cell profiles are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing maintenance hemodialysis
* Confirmed severe acute respiratory syndrome-coronavirus2 infection

Exclusion Criteria:

* Acute kidney injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal changes of interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), and interferon-gamma (IFN-γ) plasma levels during Covid19 in hemodialysis patients | Two-week observation period after Covid19 diagnosis
  Evaluation of circulating levels of pro and anti-inflammatory cytokines (pg/ml) at different time-points in patients treated with two different dialysis modalities
Longitudinal changes of soluble TLR4 (sTLR4) plasma levels during Covid19 in hemodialysis patients | Two-week observation period after Covid19 diagnosis
  Evaluation of circulating levels of soluble TLR4 (sTLR4, ng/ml)at different time-points in patients treated with two different dialysis modalities

SECONDARY OUTCOMES:
Longitudinal changes of cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), cluster of differentiation 19 (CD19), natural killer (NK) lymphocyte count and function during Covid19 in hemodialysis patients | Two-week observation period after Covid19 diagnosis
  Lymphocyte and immune cell profiles studied by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Viazzi, MD, Study Director — Unit of Nephrology, Dept Internal Medicine, Univerity of Genova and San Martino Hospital
Locations (2):
- Italy (2):
  - Ospedale IRCCS San Martino, Genova
  - Policlinico IRCCS Ospedale San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esposito P, Russo R, Conti N, Falqui V, Massarino F, Moriero E, Peloso G, Traverso GB, Garibotto G, Viazzi F. Management of COVID-19 in hemodialysis patients: The Genoa experience. Hemodial Int. 2020 Jul;24(3):423-427. doi: 10.1111/hdi.12837. Epub 2020 May 12. No abstract available. PMID 32365278
- [Background] Russo E, Esposito P, Taramasso L, Magnasco L, Saio M, Briano F, Russo C, Dettori S, Vena A, Di Biagio A, Garibotto G, Bassetti M, Viazzi F; GECOVID working group. Kidney disease and all-cause mortality in patients with COVID-19 hospitalized in Genoa, Northern Italy. J Nephrol. 2021 Feb;34(1):173-183. doi: 10.1007/s40620-020-00875-1. Epub 2020 Oct 6. PMID 33025516
- [Background] Ma Y, Diao B, Lv X, Zhu J, Chen C, Liu L, Zhang S, Shen B, Wang H. Epidemiological, Clinical, and Immunological Features of a Cluster of COVID-19-Contracted Hemodialysis Patients. Kidney Int Rep. 2020 Jun 9;5(8):1333-1341. doi: 10.1016/j.ekir.2020.06.003. eCollection 2020 Aug. PMID 32775837